CLINICAL TRIAL: NCT01388231
Title: Transfer of Manualized Cognitive-Behavioral Therapy (CBT) for Social Phobia Into Clinical Practice (SophoPrax)
Brief Title: Transfer of Manualized Cognitive-Behavioral Therapy (CBT) for Social Phobia Into Clinical Practice
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Goethe University (Other); University of Göttingen (Other)
Responsible Party: Prof. Dr. Juergen Hoyer, Dresden University of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01GV1001
Record Dates: First submitted 2011-06-08; First posted 2011-07-06 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Social Phobia
Keywords: social phobia, cognitive-behavioral therapy, treatment
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manualized CBT Group (Active Comparator): The present group is comprised of clinical practitioners performing cognitive-behavioral therapy (CBT) on social phobic patients after receiving structured clinical training on the treatment of social phobia based on the Clark and Wells (1995) model.
  Interventions: Behavioral: CBT-Manualized Intervention
- CBT Group -Treatment as Usual (Active Comparator): The present group is comprised of clinical practitioners performing cognitive-behavioral therapy (CBT) on social phobic patients, while receiving no structured training in the treatment of social phobia.
  Interventions: Behavioral: CBT-Treatment as Usual

INTERVENTIONS:
Behavioral: CBT-Manualized Intervention — Cognitive-behavioral therapy (CBT) for social phobia following the Clark and Wells (1995) model of social phobia.
  Arms: Manualized CBT Group
Behavioral: CBT-Treatment as Usual — Cognitive-behavioral therapy for social phobia following no specific model.
  Arms: CBT Group -Treatment as Usual

SUMMARY:
The study aims at examining the effects of additional training in manualized cognitive-behavioral therapy (CBT) on outcome in routine psychotherapy for social phobia. The investigators will investigate how CBT, specifically the treatment procedures and manuals proposed by Clark and Wells (1995), can be transferred from controlled trials into the less structured setting of routine clinical care, and whether the health care system benefits from such developments. Private practitioners (N=36) will be randomized to one of two treatment conditions (i.e., training in manualized CBT vs. treatment as usual without specific training). The investigators plan to enroll 160 patients (80 per condition) to be able to detect differences of d=.50 between conditions at 1-beta=.80, given the drop-out rate of 25% (N=116 completers; N=58 per condition). The study is genuinely designed to promote faster and more widespread dissemination of effective interventions. The following research questions can be examined: (1) Can manualized CBT be successfully implemented into routine outpatient care? (2) Will the new methods lead to an improvement of treatment courses aned outcomes? (3) Will treatment effects in routine psychotherapeutic treatments be comparable to those of the controlled, strictly manualized treatment of the main study?

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of Social Phobia (SCID-I)
* Liebowitz Social Anxiety Inventory Scale (LSAS) equal to or greater than 30
* age between 18 and 70 years

Exclusion Criteria:

* psychotic disorder, risk of self-harm, acute substance related disorders, personality disorders except for Cluster C (SCID-II)
* organic mental disorder
* severe medical conditions
* ongoing psychotherapy or initiation
* psychopharmacological treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Severity of Social Phobia Symptoms | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  Symptom severity will be assessed via the Liebowitz Social Anxiety Scale (LSAS).

SECONDARY OUTCOMES:
Diagnostic Status of Social Phobia | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  Diagnostic status will be assessed via SCID-I.
Assessment of Symptoms of Social Anxiety (Performance Anxiety) | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  To further assess symptoms of social anxiety, the Social Phobia Anxiety Inventory (SPAI) will be used.
Assessment of Symptoms of Social Anxiety (Social Phobic Cognitions) | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  To further assess cognitive symptoms of social anxiety, the Social Phobic Cognitions Questionnaire will be used.
Assessment of a Change in Safety Behaviors in Social Anxiety | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  To further assess safety behaviors in social anxiety the Safety Behaviors Questionnaire will be used.
Assessment of Other Social Anxiety Symptoms | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  To further assess symptoms of social anxiety, the Brief Social Phobia Scale(BSPS) will be used.
Assessment of Symptoms of Depression | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  To further assess symptoms of depression, the Beck Depression Inventory (BDI), will be employed.
Assessment of Emotion Regulation | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  To assess the level of emotion regulation, the Affective Style Questionnaire (ASQ) will be employed.
Assessment of the Quality of Life | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  To assess the quality of life in patients, the Quality of Life (QoL) questionnaire will be used.
Assessment of the Times Missing from Work | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  The times missing from work will be assessed via a separate questionnaire.
Assessment of the General Level of Severity of Social Anxiety Symptoms | Data will be collected for an expected treatment period of 30 weeks in average (corresponding to an expected average of n=25 sessions), at treatment completion, at 6 and 12 months post-treatment.
  To get a global impression from the diagnosticitian on the general level of severity of social anxiety symptoms, the Clinical Global Impression scale (CGI) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Hoyer, Prof. Dr., Principal Investigator — Technische Universität Dresden
Locations (1):
- Outpatient clinical services and day clinic center Technical University Dresden (IAP-TUD), Dresden, Saxony, Germany

REFERENCES:
- [Background] Leichsenring F, Hoyer J, Beutel M, Herpertz S, Hiller W, Irle E, Joraschky P, Konig HH, de Liz TM, Nolting B, Pohlmann K, Salzer S, Schauenburg H, Stangier U, Strauss B, Subic-Wrana C, Vormfelde S, Weniger G, Willutzki U, Wiltink J, Leibing E. The social phobia psychotherapy research network. The first multicenter randomized controlled trial of psychotherapy for social phobia: rationale, methods and patient characteristics. Psychother Psychosom. 2009;78(1):35-41. doi: 10.1159/000162299. Epub 2008 Oct 14. PMID 18852500
- [Derived] Crawcour S, Leibing E, Ginzburg D, Stangier U, Wiltink J, Hoyer J. Transfer of manualized CBT for social phobia into clinical practice (SOPHO-PRAX): a study protocol for a cluster-randomized controlled trial. Trials. 2012 May 30;13:70. doi: 10.1186/1745-6215-13-70. PMID 22647314